CLINICAL TRIAL: NCT01702610
Title: Phase II Trial of Neo-adjuvant Temozolomide Prior to Combined Temozolomide and Concurrent Accelerated Hypofractionated External Beam Radiotherapy Followed by Adjuvant Temozolomide in Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, George Shenouda, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEN-08-013; MGRT01:TMZ/GBM (Other: McGill University Health Center)
Record Dates: First submitted 2012-08-22; First posted 2012-10-08 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Glioblastoma Mutliforme
MeSH Terms: interventions — Radiotherapy, Intensity-Modulated; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temozolomide, Accelerated Hypofractionated RT (Experimental): Patient will receive two weeks of neo-adjuvant Temozolomide followed by Accelerated Hypofractionated RT for a total of 20 fractions for a total of 60Gy followed by Temozolomide for 12 cycles.
  Interventions: Radiation: IMRT Technique; Radiation: IMRT and accelerated hypofractionation technique; Radiation: neo-adjuvant TMZ followed by accelerated hypofractionated EBRT; Drug: Temozolomide and Accelerated Hypofractionation RT

INTERVENTIONS:
Radiation: IMRT Technique
Radiation: IMRT and accelerated hypofractionation technique — Intervention is the technique and accelerated fractionation used to treat GBM
Radiation: neo-adjuvant TMZ followed by accelerated hypofractionated EBRT — Two weeks of neo-adjuvant TMZ followed by XRT+TMX followed by TMZ as adjuvant component
Drug: Temozolomide and Accelerated Hypofractionation RT

SUMMARY:
Patients with GBM, who were deemed ineligible for any active protocols at our centre, received accelerated hypofractionation EBRT if 60Gy/20Fx using an IMRT technique with conventional dose of concomitant and adjuvant TMX as per the STUPP's TMZ schedule. Thirty five patients, 15 females and 20 males with a median age of 63 (range 31-78) were treated with a median KPS of 90 (range 50-100). Four patients had multicentric disease at presentation. Eight patients had biopsy only while the rest had a near total resection (n=14) and partial resection (n=13) with a median follow-up of 12.1 months, the median survival was 14.4 months.

DETAILED DESCRIPTION:
In this proposal, the total cumulative dose of TMZ is unchanged as compared to the doses used in the Stupp protocol. In this proposal, the dose of TMZ is the same, with the sole difference that TMZ will be given in a neo-adjuvant setting for two weeks and then continued at the same dose concurrently with the accelerated hypofractionated EBRT delivering 60Gy in 4 weeks. The adjuvant component of TMZ remains unchanged from current standard practice.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older
* Histological confirmation of supratentorial GBM
* KPS > 60
* Neurological function 0 or 1
* Adequate bone marrow as defined below:
* absolute neutrophil count (ANC) > 1500 cells/mm3
* platelets > 100,000 cells/mm3
* hemoglobin > 10g/dl
* Adequate renal function as defined below:
* BUN < 25mg/dl within 14 days prior to study registration
* creatinine of 63 to 103 umol/L within 14 days prior to study registration
* Adequate hepatic function as defined below:
* Bilirubin of 3 to 21 umol/L within 14 days prior to study registration
* ALT & AST < 3xnormal range within 14 days prior to study registration
* Neoadjuvant TMZ to start within 3 weeks of surgery/biopsy if no resection was deemed feasible
* A diagnostic contrast-enhanced MRI or CT scan of the brain must be performed preoperatively and postoperatively.
* History, physical and neurological examination within 14 days prior to study registration.
* For females of child-bearing potential, negative pregnancy test within 72 hours prior to starting TMZ.
* Able to sign an informed study-specific consent

Exclusion Criteria:

* Margin of contrast-enhanced residual mass closer than 15mm from the optic chiasm or optic nerves.
* Prior invasive malignancy, unless disease-free for >3years
* Recurrent or multifocal GBM
* Severe co-morbidities such as
* unstable angina
* transmural myocardial infarction within 6 months
* COPD at the time of registration
* Hepatic insufficiency
* Bacterial or fungal infection requiring IV antibiotics at the time of registration
* Acquired Immune Deficiency Syndrome (AIDS)
* Major medical illnesses or psychiatric impairments
* Pregnant women or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Percent of patients completing the study treatment | At one year
  To determine overall survival.
To assess toxicity of the regimen | At one year
  Toxicity will be assessed and graded according to CTCAE-V3

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Shenouda G, Souhami L, Petrecca K, Owen S, Panet-Raymond V, Guiot MC, Corredor AG, Abdulkarim B. A Phase 2 Trial of Neoadjuvant Temozolomide Followed by Hypofractionated Accelerated Radiation Therapy With Concurrent and Adjuvant Temozolomide for Patients With Glioblastoma. Int J Radiat Oncol Biol Phys. 2017 Mar 1;97(3):487-494. doi: 10.1016/j.ijrobp.2016.11.006. Epub 2016 Nov 15. PMID 28011051